CLINICAL TRIAL: NCT03855241
Title: Disposal Interventions for Safe Prescription Opioid Surplus Elimination: The DISPOSE Trial
Brief Title: Safely Disposing of Surplus Prescription Opioids
Acronym: DISPOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00205030
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Opioid Use
Keywords: Leftover opioids; Unused opioids; Safe prescription opioid disposal; Drug disposal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are unaware of treatment assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Informational Sheet (Active Comparator): Persons picking up an opioid prescription will receive an informational sheet that describes how to properly dispose of leftover opioid medications
  Interventions: Behavioral: Informational Sheet
- Drug Disposal Kit (Active Comparator): Persons picking up an opioid prescription will receive a drug disposal kit (DisposeRx Drug Disposal kit) and instructions on how to use it
  Interventions: Behavioral: Informational Sheet; Behavioral: DisposeRx Drug Disposal kit
- No intervention (No Intervention): Persons picking up an opioid prescription will receive no additional information or materials on disposal.

INTERVENTIONS:
Behavioral: Informational Sheet — The informational sheet details how use opioid medicines safely, and lists ways to properly dispose of leftover opioids
  Arms: Drug Disposal Kit; Informational Sheet
Behavioral: DisposeRx Drug Disposal kit — DisposeRx is a powder that is activated with water and traps leftover drugs (i.e. pills, capsules, caplets, liquids or tablets) in a semi-solid gel. The trapped drug cannot be retrieved from the resulting gel material for misuse, abuse or to leach into landfills. The participant can then throw away the biodegradable solid material in the prescription bottle into the trash, as it is safe for the environment.
  Arms: Drug Disposal Kit

SUMMARY:
This study evaluates two interventions intended to increase the safe disposal of leftover prescription opioids, compared to no intervention. Participants will receive an informational sheet describing how to safely dispose of leftover prescription opioids, an informational sheet with a drug disposal kit, or no intervention. Participants will be randomized by day for pragmatic reasons.

DETAILED DESCRIPTION:
Many persons who receive a prescription for opioids report having leftover opioids once the prescription is finished. Leftover prescription opioids serve as a reservoir of products for misuse, given 90% of people who misuse prescription opioids report obtaining the opioids from a friend, family member, or a legitimate prescription. The best way to increase the rate of safe disposal of leftover opioids is unclear. The present study will generate evidence comparing how well a drug disposal system compares with providing an informational handout on properly disposing of leftover prescription opioids. Participants will be randomized by day to one of two disposal interventions or no disposal intervention. Disposal interventions include a drug disposal kit or an informational sheet describing how to safely dispose of leftover prescription opioids. Storage and disposal characteristics for leftover prescription opioids will be measured using standardized telephone calls with participants at 3 weeks after filling the opioid prescription. If therapy is not concluded at 3 weeks or participants are not available, then a second standardized telephone call with participants will take place at 6 weeks after filling the opioid prescription.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (age ≥ 18 years) who pick up a prescription for themselves or a family member at a Johns Hopkins pharmacy
* English speaking
* Residential address and phone number in the United States
* Filling a new prescription consisting of an immediate release opioid medication (i.e., immediate release morphine, oxycodone, hydromorphone, hydrocodone, tramadol; alone or in combination with acetaminophen) with ≤ 7 days' supply

Exclusion Criteria:

* Age < 18 years
* Non-English speaking
* Residential address and/or phone number outside the United States
* Opioid medication listed in participant's active medication list prior to prescription fill
* Filling any prescription consisting of any opioid with 8 or more days' supply
* Filling any prescription consisting of any extended-release / long-acting opioid medication (i.e., extended-release morphine, oxymorphone, oxycodone, hydromorphone, fentanyl, methadone, buprenorphine)
* Filling an opioid prescription indicated for cough or shortness of breath

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Number of participants using a safe drug disposal method for leftover prescription opioids | Up to 6 weeks after prescription fill
  Participants who report "yes" to disposing of leftover prescription opioid medication using a disposal intervention that aligns with recommendations from the Food and Drug Administration (i.e., using a take-back program, drug disposal kit, or flushing in the toilet)

SECONDARY OUTCOMES:
Number of participants using any drug disposal method for leftover prescription opioids | Up to 6 weeks after prescription fill
  Participants who report "yes" to disposing of leftover prescription opioid medication using any method
Number of participants with safe storage of prescription opioids | Up to 6 weeks after prescription fill
  Participants who report "yes" to safely storing prescription opioid medication (i.e., in a locked location)
Number of participants who completed prescription opioid therapy | Up to 6 weeks after prescription fill
  Participants who report "yes" to completing therapy for prescription opioid medication

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bicket, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital/Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bicket MC, Long JJ, Pronovost PJ, Alexander GC, Wu CL. Prescription Opioid Analgesics Commonly Unused After Surgery: A Systematic Review. JAMA Surg. 2017 Nov 1;152(11):1066-1071. doi: 10.1001/jamasurg.2017.0831. PMID 28768328
- [Background] Maughan BC, Hersh EV, Shofer FS, Wanner KJ, Archer E, Carrasco LR, Rhodes KV. Unused opioid analgesics and drug disposal following outpatient dental surgery: A randomized controlled trial. Drug Alcohol Depend. 2016 Nov 1;168:328-334. doi: 10.1016/j.drugalcdep.2016.08.016. Epub 2016 Sep 20. PMID 27663358
- [Background] Rose P, Sakai J, Argue R, Froehlich K, Tang R. Opioid information pamphlet increases postoperative opioid disposal rates: a before versus after quality improvement study. Can J Anaesth. 2016 Jan;63(1):31-7. doi: 10.1007/s12630-015-0502-0. Epub 2015 Oct 2. PMID 26431852
- [Derived] Bicket MC, Fu D, Swarthout MD, White E, Nesbit SA, Monitto CL. Effect of Drug Disposal Kits and Fact Sheets on Elimination of Leftover Prescription Opioids: The DISPOSE Multi-Arm Randomized Controlled Trial. Pain Med. 2021 Apr 20;22(4):961-969. doi: 10.1093/pm/pnaa431. PMID 33576394
- See also: Provisional Drug Overdose Death Counts — https://www.cdc.gov/nchs/nvss/vsrr/drug-overdose-data.htm
- See also: Key Substance Use and Mental Health Indicators in the United States: Results from the 2017 National Survey on Drug Use and Health — https://www.samhsa.gov/data/sites/default/files/cbhsq-reports/NSDUHFFR2017/NSDUHFFR2017.htm

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT03855241/Prot_SAP_000.pdf